CLINICAL TRIAL: NCT06117007
Title: A Randomised, Placebo-controlled, Crossover Study of the Effects of a Betalain-rich Extract on Vascular Function, Sleep and Quality of Life in Middle-Aged Individuals
Brief Title: Effects of Betalains on Cardiovascular Health and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: VDF FutureCeuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HeartBeet Study
Record Dates: First submitted 2023-10-11; First posted 2023-11-03 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2023-10

CONDITIONS: Vascular Stiffness; Vasodilation; Sleep; Quality of Life
Keywords: betalains; beetroot; vascular health; sleep; quality of life
MeSH Terms: conditions — Aneurysm | interventions — Betalains

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Betalains then placebo (Experimental): Daily consumption of 1 betalain capsule (25 mg betalains) for 28 days, then crossing over to the placebo
  Interventions: Dietary Supplement: Betalains; Other: Placebo
- Placebo then betalains (Experimental): Daily consumption of 1 placebo capsule (0 mg betalains) for 28 days, then crossing over to the betalains
  Interventions: Dietary Supplement: Betalains; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Betalains — Betalains extracted from red beetroot (Beta vulgaris) encapsulated in edible capsules.
  (25 mg betalains per capsule)
Other: Placebo — Placebo capsules containing rice hulls. (0 mg betalains per capsule)

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, cross-over trial is to investigate the effects of beetroot-derived betalains on cardiovascular health, sleep and quality of life in healthy middle-aged individuals. The main question[s] it aims to answer are:

* Do betalains improve vascular function?
* Do betalains improve sleep?
* Do betalains improve quality of life?

Participants will be involved with the following:

* Consuming a daily betalain-rich or placebo capsule for a month
* Non-invasive cardiovascular measurements
* Wearing a fitness tracker for tracking physical activity and sleep
* Answering questionnaires regarding quality of life

Researchers will compare results between the intervention versus the placebo group to see if any of the study outcomes are significantly different.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 and 65 years
* BMI between 25-29.9 kg/m2
* Own a smartphone.
* Able to understand the nature of the study and give informed consent
* Have not gained or lost more than 10% of body weight (within the past 3 months)
* Not currently involved or have participated in another biomedical study (within the last 3 months)

Exclusion Criteria:

* Smoking or vaping (within the last 2 years)
* Vegetarian or vegan (due to capsule material)
* Medical history of chronic disease [coronary artery disease, previous myocardial infarction (heart attack), stroke, peripheral artery disease, diabetes mellitus, chronic kidney disease, metabolic syndrome, malignancies, etc]
* Grade II hypertension (blood pressure: >160/100 mmHg)
* Under medication that can affect the cardiovascular system (within the last 2 months)
* Taking supplements (except vitamin D and iron) (within the last month)
* Intolerances or allergies toward beetroots, dragon fruit or rice hulls
* History of excess alcohol intake or substance abuse.
* Pregnant or planning to become pregnant in the next 6 months
* Under hormonal replacement therapy (contraceptives are allowed)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Changes in flow mediated dilation (FMD) of the brachial artery | Baseline & 4 weeks
  Determine changes in flow-mediated dilation (FMD) of the brachial artery after 4 weeks consumption of 25 mg betalains

SECONDARY OUTCOMES:
Changes in flow mediated dilation (FMD) of the brachial artery | Baseline & 90 minutes
  Determine changes in flow-mediated dilation (FMD) of the brachial artery at 90 minutes after consumption of 25 mg betalains
Changes in blood pressure | Baseline, 90 minutes and 4 weeks
  Determine changes in systolic and diastolic blood pressure at 90 minutes and 4 weeks after consumption of 25 mg betalains
Changes in arterial stiffness | Baseline and 4 weeks
  Determine changes in pulse-wave velocity and pulse-wave analysis after 4 weeks of consumption of 25 mg betalains using applanation tonometry on SphygmoCor system.
Changes in heart rate | Baseline, 90 minutes and 4 weeks
  Determine changes in heart rate at 90 minutes and 4 weeks after consumption of 25 mg betalains
Changes in sleep quality (sleep duration, percent of light, deep and REM sleep and etc.) | Baseline and 4 weeks
  Determine changes in sleep quality (sleep duration, percent of light, deep and REM sleep etc.) after 4 weeks of consumption of 25 mg betalains using wearable activity tracker.
Changes in quality of life (quality of life scores and physical activity) | Baseline and 4 weeks
  Determine changes in quality of life after 4 weeks consumption of 25 mg betalains via WHOQoL-100 questionnaire, Short Form-36 (SF-36) survey, and physical activity on wearable activity tracker.
Changes in blood flow velocity | Baseline, 90 minutes and 4 weeks
  Determine changes in blood flow velocity at 90 minutes and 4 weeks after consumption of 25 mg betalains

OTHER OUTCOMES:
Changes in plasma erythropoietin | Baseline, 90 minutes and 4 weeks
  Determine changes in plasma erythropoietin at 90 minutes and 4 weeks after consumption of 25 mg betalains
Changes in red blood cell deformability | Baseline, 90 minutes and 4 weeks
  Determine changes in red blood cell deformability at 90 minutes and 4 weeks after consumption of 25 mg betalains measured via osmotic gradient ektacytometry.
Plasma betalains and polyphenol metabolites | Baseline, 90 minutes and 4 weeks
  Measured by liquid chromotography-mass spectrometry (LC/MS) post-consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — King's College London
Locations (1):
- Metabolic Research Unit (King's College London), London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No